CLINICAL TRIAL: NCT03141580
Title: Long-term Follow-up Near-infrared Spectroscopy and Intravascular Ultrasound Imaging of Internal Carotid Artery Stenosis Treated With Stenting
Brief Title: Long-term Follow-up NIRS-IVUS Imaging of Pre-existing Carotid Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Collaborators: professor Josef Veselka (Unknown); associate professor Petr Hájek (Unknown); Martin Horváth (Unknown)
Responsible Party: Principal Investigator, Cyril štěchovský, Principal Investigator, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK-953/16
Record Dates: First submitted 2017-04-03; First posted 2017-05-05 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Carotid Atherosclerosis; Carotid Artery Stenting; Atherosclerotic Plaque; Near Infrared Spectroscopy; Restenosis
MeSH Terms: conditions — Carotid Artery Diseases; Plaque, Atherosclerotic | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Subjects with carotid stent who consented to undergo near-infrared spectroscopy and intravascular ultrasound imaging.
  Interventions: Diagnostic Test: Near-infrared spectroscopy and intravascular ultrasound (NIRS-IVUS)

INTERVENTIONS:
Diagnostic Test: Near-infrared spectroscopy and intravascular ultrasound (NIRS-IVUS) — Examination of the extracranial portion of the internal and common carotid artery with pre-existing stent with NIRS-IVUS.

SUMMARY:
The 'Long-term Follow-up Near-infrared Spectroscopy and Intravascular Ultrasound Imaging of Internal Carotid Artery Stenosis Treated With Stenting' trial is an academic research project. It follows already published results of a research on carotid plaque composition in patients undergoing carotid stenting.

Patients who were treated with carotid stenting will be invited to participate on the trial. The written informed consent will be needed. The participants will undergo carotid angiography, intravascular near-infrared spectroscopy and intravascular ultrasound of the extracranial portion of the internal and common carotid artery with implanted stent.

The aim of the trial is to describe long-term change of the luminal and stent dimensions, vessel wall remodeling and plaque composition after carotid stenting. The findings will help to understand the long-term effect of carotid stenting on the carotid stenosis and mechanisms of plaque stabilization - sealing with stent.

ELIGIBILITY:
Inclusion Criteria:

* previous carotid stenting
* data from periprocedural NIRS-IVUS available
* written informed consent

Exclusion Criteria:

* occlusion of the carotid artery on the side of the implanted stent
* indication for carotid intervention on the side of the implanted stent
* high procedural risk (difficult anatomy, risk of puncture site bleeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Temporal change of lipid core burden index (LCBI) | 16 months
  Difference between LCBI (a dimensionless number) within the segment of the carotid artery with implanted stent in the time point of the carotid stenting (baseline LCBI) and in the time point of study intervention (follow-up LCBI). Data from NIRS.

SECONDARY OUTCOMES:
Late lumen change | 16 months
  Difference between luminal volume (mm3) within the segment of the carotid artery with implanted stent in the time point of the carotid stenting (baseline lumen volume) and in the time point of study intervention (follow-up lumen volume). Data from IVUS.
Late stent expansion | 16 months
  Difference between stent volume (mm3) within the segment of the carotid artery with implanted stent in the time point of the carotid stenting (baseline stent volume) and in the time point of study intervention (follow-up stent volume). Data from IVUS.

CONTACTS AND LOCATIONS:
Locations (1):
- Motol University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stechovsky C, Hajek P, Horvath M, Spacek M, Veselka J. Near-infrared spectroscopy combined with intravascular ultrasound in carotid arteries. Int J Cardiovasc Imaging. 2016 Jan;32(1):181-8. doi: 10.1007/s10554-015-0687-x. Epub 2015 Jun 5. PMID 26044524
- [Background] Stechovsky C, Hajek P, Horvath M, Spacek M, Veselka J. Composition of carotid artery stenosis and restenosis: A series of patients assessed with intravascular ultrasound and near-infrared spectroscopy. Int J Cardiol. 2016 Mar 15;207:64-6. doi: 10.1016/j.ijcard.2016.01.104. Epub 2016 Jan 9. No abstract available. PMID 26797333
- [Background] Horvath M, Hajek P, Muller JE, Honek J, Stechovsky C, Spacek M, Veselka J. First-in-man near-infrared spectroscopy proof of lipid-core embolization during carotid artery stenting. Arch Med Sci. 2016 Aug 1;12(4):915-8. doi: 10.5114/aoms.2016.60974. Epub 2016 Jul 1. No abstract available. PMID 27478475
- [Background] Horvath M, Hajek P, Stechovsky C, Honek J, Spacek M, Veselka J. The role of near-infrared spectroscopy in the detection of vulnerable atherosclerotic plaques. Arch Med Sci. 2016 Dec 1;12(6):1308-1316. doi: 10.5114/aoms.2016.62904. Epub 2016 Oct 24. PMID 27904523
- [Background] Horvath M, Hajek P, Stechovsky C, Honek J, Veselka J. Intravascular Near-Infrared Spectroscopy: A Possible Tool for Optimizing the Management of Carotid Artery Disease. Int J Angiol. 2015 Sep;24(3):198-204. doi: 10.1055/s-0035-1558644. Epub 2015 Aug 6. PMID 26417188
- [Background] Veselka J, Spacek M, Hajek P, Horvath M, Stechovsky C, Zimolova P. Impact of single versus double vessel carotid disease on long-term survival in patients treated with carotid stenting. Int J Cardiol. 2014 Oct 20;176(3):1299-300. doi: 10.1016/j.ijcard.2014.07.165. Epub 2014 Aug 3. No abstract available. PMID 25127969
- [Background] Veselka J, Spacek M, Horvath M, Stechovsky C, Homolova I, Zimolova P, Hajek P. Impact of coexisting multivessel coronary artery disease on short-term outcomes and long-term survival of patients treated with carotid stenting. Arch Med Sci. 2016 Aug 1;12(4):760-5. doi: 10.5114/aoms.2016.60964. Epub 2016 Jul 1. PMID 27478456
- [Background] Spacek M, Zimolova P, Veselka J. Carotid artery stenting without post-dilation. J Interv Cardiol. 2012 Apr;25(2):190-6. doi: 10.1111/j.1540-8183.2011.00694.x. Epub 2011 Dec 8. PMID 22150803
- [Background] Spacek M, Martinkovicova L, Zimolova P, Veselka J. Mid-term outcomes of carotid artery stenting in patients with angiographic string sign. Catheter Cardiovasc Interv. 2012 Jan 1;79(1):174-9. doi: 10.1002/ccd.23144. Epub 2011 Nov 30. PMID 21542110
- [Background] Veselka J, Cerna D, Zimolova P, Martinkovicova L, Fiedler J, Hajek P, Maly M, Zemanek D, Duchonova R. Feasibility, safety, and early outcomes of direct carotid artery stent implantation with use of the FilterWire EZ Embolic Protection System. Catheter Cardiovasc Interv. 2009 May 1;73(6):733-8. doi: 10.1002/ccd.21936. PMID 19198010
- [Background] Veselka J, Cerna D, Zimolova P, Blasko P, Fiedler J, Hajek P, Maly M, Zemanek D, Duchonova R. Thirty-day outcomes of direct carotid artery stenting with cerebral protection in high-risk patients. Circ J. 2007 Sep;71(9):1468-72. doi: 10.1253/circj.71.1468. PMID 17721030
- [Background] Stechovsky C, Hajek P, Horvath M, Veselka J. Effect of stenting on the near-infrared spectroscopy-derived lipid core burden index of carotid artery plaque. EuroIntervention. 2019 Jun 12;15(3):e289-e296. doi: 10.4244/EIJ-D-17-01054. PMID 29957596
- [Derived] Stechovsky C, Hajek P, Roland R, Horvath M, Veselka J. Long-term changes after carotid stenting assessed by intravascular ultrasound and near-infrared spectroscopy. Cardiovasc Diagn Ther. 2021 Dec;11(6):1180-1189. doi: 10.21037/cdt-21-160. PMID 35070788